CLINICAL TRIAL: NCT06196788
Title: Gemcitabine and Nab-paclitaxel Venous Injection Plus Transcatheter Arterial Infusion to Patients With Advanced Pancreatic Cancer
Brief Title: Transcatheter Arterial Infusion to Patients With Advanced Pancreatic Cancer
Acronym: PTCA199-9
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Guopei Luo, Professor, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PTCA199-9
Record Dates: First submitted 2023-12-26; First posted 2024-01-09 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2024-03

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Gemcitabine; Taxes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- gemcitabine and nab-paclitaxel venous injection plus transcatheter arterial infusion (Experimental): nab-paclitaxel (120 mg per square meter of body-surface area) followed by gemcitabine (1000 mg per square meter) on days 1 (venous injection), 8 (venous injection), and 15 (transcatheter arterial infusion) every 4 weeks.
  Interventions: Drug: Gemcitabine; Drug: Nab paclitaxel

INTERVENTIONS:
Drug: Gemcitabine — 1000 mg per square meter
Drug: Nab paclitaxel — 120 mg per square meter of body-surface area

SUMMARY:
The purpose of this study is to evaluate the efficacy of gemcitabine and nab-paclitaxel venous injection plus transcatheter arterial infusion to Patients with Advanced Pancreatic Cancer.

DETAILED DESCRIPTION:
Pancreatic cancer is a highly lethal malignancy with a 5-year survival less than 10%. Approximately 80% of patients with pancreatic cancer are diagnosed at an advanced stage. Chemotherapy is one of the major treatments for advanced pancreatic cancer. The MPACT trial has confirmed the efficacy of gemcitabine combined with nab-paclitaxel as the first-line treatment to metastatic pancreatic cancer. However, the side-effects related to gemcitabine combined with nab-paclitaxel including anemia, hand/foot numbness, fatigue, nausea, and malnutrition have impaired the tolerability of the regimen.

Regional intra-arterial infusion chemotherapy helps to deliver anticancer drugs into the carcinoma tissue more selectively and is considered to be a potential alternative treatment for advanced pancreatic adenocarcinoma with less systemic adverse effects. Ohigashi et al first reported that intraarterial chemotherapy using 5-fluorouracil improved the prognosis and quality of life in patients with advanced pancreatic carcinoma.

The purpose of this study is to evaluate the efficacy of gemcitabine and nab-paclitaxel venous injection plus transcatheter arterial infusion to patients with advanced pancreatic cancer. Progression-free survival (PFS), objective response rate (ORR), overall survival (OS) and disease control rate (DCR) are measured every three weeks.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand and the willingness to sign a written informed consent document.
* Age ≥ 18 years and ≤ 80 years.
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2.
* Histologically or cytologically confirmed advanced pancreas adenocarcinoma.
* Primary pancreatic cancer without major anti-cancer treatments.
* Locally advanced, or metastatic pancreatic cancer.
* Presence of at least of one measurable lesion in agreement to RECIST criteria.
* The expected survival ≥ 3 months.
* Adequate organ performance based on laboratory blood tests.
* Patients who are willing or able to comply with study procedures.

Exclusion Criteria:

* Pregnant or nursing women.
* Patients who have received anti-tumor chemotherapy, radiotherapy, or other treatments.
* The diagnosis was confirmed by pathology as non-adenocarcinoma of pancreas.
* Inflammation of the digestive tract, including pancreatitis, cholecystitis, cholangitis, etc.
* Severe and uncontrollable accompanying diseases that may affect protocol compliance or interfere with the interpretation of results.
* Cardiovascular and cerebrovascular accidents.
* Allergic to study drugs.
* Other serious accompanying illnesses, which, in the researcher's opinion, could seriously adversely affect the safety of the treatment.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Overall survival，OS | At the end of Cycle 1 (each cycle is 28 days)
  OS of subjects from recruiting to the time of death from any cause

SECONDARY OUTCOMES:
progression-free survival, PFS | At the end of Cycle 1 (each cycle is 28 days)
  PFS of subjects from recruiting to the time of disease progression
objective response rate (ORR), | At the end of Cycle 1 (each cycle is 28 days)
  CR + PR
disease control rate (DCR) | At the end of Cycle 1 (each cycle is 28 days)
  CR + PR + SD

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Aigner KR, Gailhofer S, Selak E, Aigner K. Intra-arterial infusion chemotherapy versus isolated upper abdominal perfusion for advanced pancreatic cancer: a retrospective cohort study on 454 patients. J Cancer Res Clin Oncol. 2019 Nov;145(11):2855-2862. doi: 10.1007/s00432-019-03019-6. Epub 2019 Sep 10. PMID 31506738
- [Background] Liu X, Yang X, Zhou G, Chen Y, Li C, Wang X. Gemcitabine-Based Regional Intra-Arterial Infusion Chemotherapy in Patients With Advanced Pancreatic Adenocarcinoma. Medicine (Baltimore). 2016 Mar;95(11):e3098. doi: 10.1097/MD.0000000000003098. PMID 26986149
- [Background] Endo S, Kawaguchi S, Terada S, Shirane N. Hepatic Arterial Infusion Chemotherapy for Liver Metastases Following Standard Chemotherapy for Pancreatic Cancer. Intern Med. 2021 Jan 15;60(2):223-229. doi: 10.2169/internalmedicine.5449-20. Epub 2020 Sep 19. PMID 32963157
- [Background] Qiu B, Zhang X, Tsauo J, Zhao H, Gong T, Li J, Li X. Transcatheter arterial infusion for pancreatic cancer: a 10-year National Cancer Center experience in 115 patients and literature review. Abdom Radiol (NY). 2019 Aug;44(8):2801-2808. doi: 10.1007/s00261-019-02022-2. PMID 31025067